CLINICAL TRIAL: NCT04109950
Title: An Open-label Extension Study to Assess the Safety and Tolerability of SEP-363856 in Subjects With Schizophrenia
Brief Title: A Clinical Study to Evaluate the Long-term Safety and Tolerability of an Investigational Drug in People With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early, main goals achieved
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-303; 2019-000696-16 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: This is a 52-week, outpatient, multicenter, flexible-dose, open-label extension study designed to evaluate the long-term safety and tolerability of SEP-363856 (25 to 100 mg/day) for treatment of participants with schizophrenia who have completed Treatment Period of one of two following double-blind studies: Study SEP361-301 (NCT04072354) or Study SEP361-302 (NCT04092686).
  The study will consist of two periods: An Open-Label Extension (OLE) Treatment Period (up to 52 weeks); and a Follow-up visit at 7±2 days after last study drug dose for participants who complete the Treatment Period & those who prematurely discontinue from study.
  The adolescent cohort includes participants who were 13 to 17 years of age, at time of consent in the SEP361-301 study. For adolescent participants, a reliable informant (e.g., parent, legal guardian, or caregiver) of participant should accompany participant at each visit and support and monitor the participants compliance with taking study medication.
Masking Description: open - label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental): SEP-363856 25mg, 50mg, 75mg, 100mg flexibly dosed once daily
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 25mg, 50mg, 75mg, 100mg tablet flexibly dosed once daily

SUMMARY:
This is a clinical trial to determine the long-term safety and tolerability of an investigational drug in people with schizophrenia. Participants in the study will receive the drug being studied. This study is accepting male and female participants between 13 and 65 years old who have been diagnosed with schizophrenia and have completed Study SEP361-301 (NCT04072354) or Study SEP361-302 (NCT04092686). This study will be conducted in approximately 80 study centers worldwide. The treatment duration for this study is one (1) year.

DETAILED DESCRIPTION:
An open-label extension study to assess the safety and tolerability of SEP-363856 in participants with schizophrenia This is an open-label extension study to evaluate long-term safety and tolerability of SEP-363856. This is a 52-week, outpatient, multicenter, flexible-dose, open-label extension study designed to evaluate the long-term safety and tolerability of SEP-363856 (25 to 100 mg/day) for the treatment of participants with schizophrenia who have completed the Treatment Period of one of the two following double-blind studies: Study SEP361-301 (NCT04072354) or Study SEP361-302 (NCT04092686).

Sumitomo Pharma America Inc. was the former Sponsor and conducted this study. Sumitomo was responsible for analysis and clinical study report (CSR) completion. Otsuka took over study after IND was transferred and is concluding activities with registry postings.

ELIGIBILITY:
Inclusion Criteria:

1. Participant (or participants parent/legal guardian for adolescents) must give written informed consent and privacy authorization prior to participation in the study; adolescents must also provide informed assent.
2. Participant has completed the Treatment Period of Study SEP361-301 or Study SEP361-302.
3. Participant has not taken any medication other than the study drug and protocol-allowed medications for the purpose of controlling schizophrenia symptoms during Study SEP361-301 or SEP361-302.
4. Female participant must have a negative urine pregnancy test at the End of Treatment (EOT) Visit of Study SEP361-301 or Study SEP361-302.
5. Female participants of childbearing potential must agree to use highly effective and reliable contraception throughout the study and for at least 30 days after the last dose of study drug has been taken.
6. Male participants must agree to avoid fathering a child and use highly effective methods of birth control from screening in Study SEP361-301 or Study SEP361-302, until at least 30 days after the last study drug administration in the present study (SEP361-303).

Exclusion Criteria

1. Participant answered "yes" to "suicidal ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the Columbia Suicide Severity Rating Scale (C-SSRS) assessment at the End of treatment (EO) Visit of Study SEP361-301 or SEP361-302.
2. Participant has a clinically significant abnormality including physical examination, vital signs, ECG, or laboratory test at the EOT Visit of Study SEP361-301 or SEP361-302 that the investigator in consultation with the medical monitor considers to be inappropriate to allow participation in the study.
3. Participant has a positive urine drug screen (UDS) at the EOT Visit of Study SEP361-301 or SEP361-302. However, a positive UDS test may not result in exclusion of participants if the Investigator determines that the positive test is as a result of prescription medicine(s). participants may enter this study before the urine drug screen results are received from the central laboratory. However, after receipt and review of the results any participant meeting this exclusion criterion must be discontinued from the study. Retesting of the UDS is allowed once with prior approval from the Medical Monitor with the retest used to determine eligibility
4. Female participant is pregnant or lactating.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
The incidence of overall Adverse Events (AEs), Serious Adverse Events (AEs), and Adverse Events (AEs) leading to discontinuation | 53 Weeks

CONTACTS AND LOCATIONS:
Locations (61):
- United States (22):
  - Research Site, Little Rock, Arkansas
  - Research Site, Rogers, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Culver City, California
  - Research Site, Lemon Grove, California
  - Research Site, Long Beach, California
  - Research Site, Montclair, California
  - Research Site, San Diego, California
  - Research Site, Sherman Oaks, California
  - Research Site, Miami Springs, Florida
  - Research Site, Oakland Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Lake Charles, Louisiana
  - Research Site, Gaithersburg, Maryland
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Marlton, New Jersey
  - Research Site, New York, New York
  - Research Site, Dayton, Ohio
  - Research Site, Austin, Texas
  - Research Site, Richardson, Texas
- Bulgaria (8):
  - Research Site, Burgas
  - Research Site, Kardzhali
  - Research Site, Novi Iskar
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
- Colombia (2):
  - Research Site, Barranquilla
  - Research Site, Bogotá
- Research Site, Zagreb, Croatia
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Riga
  - Research Site, Strenči
- Russia (9):
  - Research Site, Chelyabinsk
  - Research Site, Matrosy
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Stavropol
  - Research Site, Talagi
- Serbia (8):
  - Research Site, Belgrade
  - Research Site, Gornja Toponica
  - Research Site, Kovin
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Kneževac
  - Research Site, Novi Sad
  - Research Site, Vršac
- Ukraine (8):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Nove
  - Research Site, Odesa
  - Research Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com